CLINICAL TRIAL: NCT04455555
Title: Efficacy and Safety of Rotigotine in the Treatment of Patients With Early Stage of Primary Parkinson's Disease
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Peking University Third Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: PUTH2018083
Record Dates: First submitted 2020-06-28; First posted 2020-07-02 (Actual); Last update posted 2020-07-02 (Actual); Status verified 2020-07

CONDITIONS: Parkinson's Disease
Keywords: Parkinson's disease；rotigotine
MeSH Terms: conditions — Parkinson Disease

STUDY DESIGN:
Who Masked: Participant, Investigator
Masking Description: participant and investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- rotigotine treatment group (Experimental): rotigotine sustained release microspheres therapy by injection
  Interventions: Drug: LY03003( the name of rotigotine)
- placebo comparator (Placebo Comparator): placebo comparator/null microspheres
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: LY03003( the name of rotigotine) — LY03003 (Continuous Dopamine Stimulation) sustained release microspheres / injection once a week 4 weeks followed by 24 weeks until 28 weeks.
  Arms: rotigotine treatment group
Other: Placebo — Null sustained release microspheres placebo / injection once a week 4 weeks followed by 24 weeks until 28 weeks.
  Arms: placebo comparator

SUMMARY:
The efficacy and safety of rotigotine in the treatment of patients with early stage of primary Parkinson's disease

DETAILED DESCRIPTION:
To evaluate the efficacy and safety of rotigotine sustained release microspheres therapy by injection in the treatment of patients with early stage of primary Parkinson's disease

ELIGIBILITY:
Inclusion Criteria:

* Subjects or their legal representatives understand and wish to participate in this clinical study and voluntarily sign the informed consent dated;
* In the investigator's judgment, believe that the subject or his legal representative is trustworthy and able to comply with the study protocol, visit plan, or receive the study drug treatment as required;
* During screening (interview 1) The subjects were older than 30 years old, regardless of gender;
* The subject had primary Parkinson's disease for 55 years and was diagnosed based on major signs such as delayed movement and at least one of the following symptoms: quiescence tremor, rigidity or postural reflexes, and no other known or suspected cause of Parkinson's disease;
* Hoehn-yahr stage 3 in the "open" state (excluding phase 0);
* Brief mental State examination (MMSE) ≥ 25;
* At baseline (visit 2), the exercise score (Part III) of the Unified Parkinson's Disease Rating Scale (U PDRS) under the "open" condition was greater than or equal to 10;
* If the subjects are receiving anticholinergic drugs (such as benzalkonium tropic, benzene hai suo, diethyl promethazine, its organism and than pp board), monoamine oxidase B (MAO B) inhibitors, N - Methyl - d - aspartate (NMDA) antagonist (such as amantadine) treatment, must dose before baseline visit (2) is stable at least 28 days, and maintain the dose treatment during the study period;
* Childbearing age women (such as: no sterilization surgery or postmenopausal women is less than 1 year) or male subjects agreed to during the entire study (screening visit to the end of the study) and reliable contraceptive measures (birth control pills, use a condom, abstinence, etc.), and the screening visit (l) and the baseline visit (2), the childbearing age women of pregnancy test results were negative.

Exclusion Criteria:

* A history of globulin resection, thalamic destruction, deep brain stimulation or fetal tissue transplantation;
* Dementia, active mental illness or hallucinations, major depression
* Those who received dopamine agonist within 28 days before baseline (visit 2);
* Those who received levodopa preparations (including levodopa compound preparations) within 28 days before baseline (visit 2), or those who received levodopa preparations for more than 6 months after diagnosis; Patients who received any of the following drugs: amphetamine or alpha within 28 days prior to baseline (visit 2)
* Receiving Central nervous system active drug therapy (e.g., tranquilizers, sleeping pills, antidepressants, antianxiety medications), except for those who have been on a stable dose for at least 28 days prior to baseline (visit 2) and are likely to remain stable during the study period;
* Atypical Parkinson's disease symptoms caused by the use of drugs (e.g., metoclopramide, flunarizine), hereditary metabolic diseases of the nervous system (e.g., Wilson's disease), encephalitis, cerebrovascular diseases, or degenerative diseases (e.g., progressive supranuclear palsy);
* Patients with a history of epilepsy, or with a history of stroke or transient ischemic stroke within 1 year before the visit;
* Intolerance or allergy to antiemetic drugs such as domperidone, ondansetron, tropisetron, granisetron;
* Patients with clinically significant liver function abnormalities are defined as 1.5 times of the upper limit of the reference range of total bilirubin > or 2 times of the upper limit of the reference range of alanine aminotransferase (ALT) or aspartate aminotransferase (AST) >;
* Abnormal renal function with clinical significance (serum creatinine > 2.0 mg/dL);
* Uncontrolled or significant cardiovascular disease, including New York Heart Association grade 2 or above congestive heart failure, unstable angina, myocardial infarction, or arrhythmias requiring treatment at screening (visit 1) in the 6 months prior to first administration of the study drug;
* During screening (interview I);
* A history of symptomatic postural hypotension; Systolic blood pressure reduction greater than or equal to 20 MMHG or diastolic blood pressure reduction greater than or equal to 10 mmHg during screening (visit l) and baseline (visit 2) from baseline to upright position for 1 or 3 minutes; Or patients with horizontal systolic blood pressure < 105 mmHg during screening (visit I) and baseline (visit 2);
* Subjects with evidence of impulse control disorder (ICD) during screening (interview L);
* A history of suicide attempt (including actual attempt, interruption of attempt or failure of attempt) or suicidal ideation in the past 6 months, defined as "yes" to question 4 or 5 on the Columbine Suicide Severity Rating Scale (C-SSRS) at screening (interview L); those
* Patients with a history of narcolepsy;
* Screening (interview L) For those who had a history of alcohol abuse, drug abuse or drug addiction in the first 5 years, alcoholism was defined as drinking more than 14 units of alcohol per week (1 unit = 360 ml beer or 45 ml spirits with 40% alcohol or 150 ml wine);
* Screening for malignant tumors within 5 years before surgery, except adequately treated carcinoma in situ of the cervix, basal cell or squamous cell carcinoma of the skin, local prostate cancer after radical surgery, and intraductal carcinoma in situ of the breast;
* Women during pregnancy or lactation;
* Previous participants in the Rotigotine trial were intolerant or had poor efficacy;
* Allergic to or known to be allergic to rotigotine or rotigotine microsphere preparations;
* Those who have participated in other drug clinical trials within 3 months prior to screening;
* Any other medical condition, mental condition, or laboratory abnormality of clinical significance that the investigator determines may interfere with the subject's ability to participate in the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 294 (Actual)
Dates: Start 2018-08-01 (Actual); Primary Completion 2019-02-01 (Actual); Study Completion 2019-02-01 (Actual)

PRIMARY OUTCOMES:
Changes in the total Unified Parkinson Disease Rating Scale (UPDRS) (II +III) score | 32 weeks after treatment
  Changes in the total Unified Parkinson Disease Rating Scale (UPDRS) (II +III) score relative to baseline from baseline to the end of the double-blind dose maintenance period, The UPDRS scale refers to Unified Parkinson Disease Rating Scale, and it is a rating tool used to gauge the course of Parkinson's disease in patients. Some sections of the UPDRS scale require multiple grades assigned to each extremity with a possible maximum of 199 points. A score of 199 on the UPDRS scale represents the worst (total disability) with a score of zero representing (no disability).

SECONDARY OUTCOMES:
Unified Parkinson Disease Rating Scale (UPDRS) maximum table (II +III) total score | 32 weeks after treatment
  Unified Parkinson Disease Rating Scale (UPDRS) maximum table (II +III) total score relative to baseline from baseline to the end of the double-blind dose maintenance period, The UPDRS scale refers to Unified Parkinson Disease Rating Scale, and it is a rating tool used to gauge the course of Parkinson's disease in patients. Some sections of the UPDRS scale require multiple grades assigned to each extremity with a possible maximum of 199 points. A score of 199 on the UPDRS scale represents the worst (total disability) with a score of zero representing (no disability).
changes in part II of the Unified Parkinson Disease Rating Scale relative to baseline | 32 weeks after treatment
  Changes from baseline to the end of the double-blind dose maintenance period in part III of the Unified Parkinson Disease Rating Scale relative to baseline; The Unified Parkinson Disease Rating Scale scale refers to Unified Parkinson Disease Rating Scale, and it is a rating tool used to gauge the course of Parkinson's disease in patients. Some sections of the Unified Parkinson Disease Rating Scale scale require multiple grades assigned to each extremity with a possible maximum of 199 points. A score of 199 on the Unified Parkinson Disease Rating scale represents the worst (total disability) with a score of zero representing (no disability).
changes in the severity (SI) score; | 32 weeks after treatment
  From baseline to the end of the double-blind dose maintenance period, changes in the severity (SI) score of Item 1 ;The Severity Score (ISS) scores ranges from 0 to 75 (i.e. Abbreviated Scale (AIS) scores of 6 for each injury in every body region according to its relative severity). If an injury is assigned an Abbreviated Injury Scale (AIS) of 6 (identified currently as untreatable injury or unsurvivable injury), the ISS score is automatically assigned 75. Since a score of 6 ("unsurvivable") indicates the futility of further medical care in preserving life, this may mean a cessation of further care in triage for a patient with a score of 6 in any category.
Changes in pd Questionnaire (PDQ-8) scores | 32 weeks after treatment
  Changes in pd Questionnaire (PDQ-8) scores relative to baseline from baseline to the end of the double-blind dose maintenance period; the higher the score, the worse of life quality
Changes in pd sleep Disorders Scale (PDSS) score | 32 weeks after treatment
  Changes in pd sleep Disorders Scale (PDSS) score from baseline to the end of the double-blind dose maintenance period. The overall PDSS is the summary score of the single PDSS items. If the single items have values between 0 (= worst case) to 10 (= best case) the total score can range between 0 and 150. Score 150 means the best case.
Changes in Beck Depression Inventory II (BDI-II) scores | 32 weeks after treatment
  Changes in Beck Depression Inventory II (BDI-II) scores relative to baseline from baseline to the end of the double-blind dose maintenance period. Each item of the BDI-II is rated along a 4-point Likert scale from 0 to 3； Items are summed to produce a total score（0-63） with higher scores representing more depressive symptoms.

CONTACTS AND LOCATIONS:
Overall Officials: Dongsheng Fan, MD.PHD, Principal Investigator — Peking University Third Hospital
Locations (1):
- Peking University Third Hospital, Beijing, China

IPD SHARING:
Plan to Share IPD: No